CLINICAL TRIAL: NCT04274712
Title: Non-invasive Test for Acute Rejection Identification in Heart Transplanted Patients: a Pilot Retrospective Study
Brief Title: Non-invasive Test for Acute Rejection Identification in Heart Transplanted Patients
Acronym: INNOGRAFTRS001
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Myway Gentics Srl (Industry)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Other Study IDs: INNOGRAFTRS001
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Acute Rejection of Cardiac Transplant
Keywords: liquid biopsy; cfDNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma from transplanted patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: INNOGRAFT Heart Suite — Liquid biopsy to identify acute rejection

SUMMARY:
Aim of the study is to test INNOGRAFT Heart Suite in a clinical setting, using a previously collected set of plasma samples from patients who underwent heart transplant and routinely or symptoms-based surveillance during the period 2016- 2019.

DETAILED DESCRIPTION:
Aim of the study is to test INNOGRAFT Heart Suite in a clinical setting, using a previously collected set of plasma samples from patients who underwent heart transplant and routinely or symptoms-based surveillance during the period 2016- 2019.

1. Primary end-point

   • To evaluate specificity and sensitivity of INNOGRAFT Heart Suite in identifying transplant rejection, using blood samples collected from heart transplanted patients during the same day of endomyocardial biopsy (EMB) using the histological study of EMB specimen as reference technique.

   We will evaluate:
   1. Presence of rejection (Yes/No),
   2. Correct classification of rejection according to ISHLT 2004 guidelines. Rejection will be considered Yes if ISHLT 2004 grading is >1R. We chose ISHLT scale because it has been previously used in studies aimed at sensitivity assessment of other techniques (Deng et al. 2006) and because changes of therapeutic protocol are usually considered in presence of rejection grade higher than 2R.
2. Secondary end-points

   * To evaluate the accuracy of INNOGRAFT Heart Suite in discriminating between the classes of rejection according to ISHLT 2004 guidelines using histological study of heart samples from EMB as reference technique
   * To look for potential clinical modifiers of cfDNA levels, as quantitatively determined through INNOGRAFT Heart Suite, for every given rejection class. Expected modifiers are inflammatory states not related to rejection and infections. We will also consider the influence of other factors such as gender, age, pregnancy, comorbidities such as other organ failure, diabetes, cancer.
   * To find if a correlation between basal donor cfDNA levels, as quantitatively determined through INNOGRAFT Heart Suite on blood samples routinely collected for surveillance or symptoms-based surveillance, and clinical outcomes exists. Clinical outcome considered will be rejection, arrythmias, graft failure, hospitalization, death.
   * To find if a correlation between donor cfDNA levels, as quantitatively determined through INNOGRAFT Heart Suite on blood samples routinely collected for surveillance or symptoms-based surveillance, and parameters of cardiac function obtained through right heart catheterization exists. Cardiac catheterization will measure cardiac index, left atrium wedge, right ventricle pressure, pulmonary artery avarage pressure.
   * To find if a correlation between donor cfDNA levels, as quantitatively determined through INNOGRAFT Heart Suite on blood samples routinely collected for surveillance or symptoms-based surveillance, and blood levels of calcineurin inhibitor/proliferation inhibitor (in therapeutic range/outside therapeutic range) exists in each patient and between patients. Calcineurin inhibitor, proliferation inhibitor and steroids are routine therapy for patients who underwent heart transplant. Blood levels are routinely measured in patient treated with calcineurin inhibitor or proliferation inhibitor protocols. The aim is to identify through cfDNA measure, the correct patient-specific level of immunosuppression.
   * To find if differences in basal donor cfDNA levels, as quantitatively determined through INNOGRAFT Heart Suite on blood samples routinely collected for surveillance or symptoms-based surveillance, between rATG-treated and rATG-untreated patients exist. rATG is intended as induction therapy protocol before heart transplant.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients must fulfill all the following inclusion criteria.

1. Age≥18 years;
2. Heart transplanted during 2016-2019 and under surveillance for preventing acute rejection;
3. Heart transplanted before 2016 but undergoing routinely or symptom-based surveillance for preventing acute rejection;
4. Signed written informed consent for reuse of biosamples for research purposes; OR Signed written informed consent for study partecipation;
5. Underwent at least 1 blood sampling at the same time of the EMB;
6. Clinical data collected during at least 1 surveillance visit (same time of blood sampling and EMB) available;
7. Availability of EMB readings for EMB performed at the same time of blood sampling.

Exclusion Criteria:

1. They were subjected to re-transplantation
2. They were subjected to multi-organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplanted consecutive adult patients , who underwent their regular surveillance protocol during the first 3 years post intervention.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Comparison with gold standard: endomyocardial biopsy | 6 months
  To evaluate specificity and sensitivity of INNOGRAFT Heart Suite in identifying transplant rejection, using blood samples collected from heart transplanted patients during the same day of endomyocardial biopsy (EMB) using the histological study of EMB specimen as reference technique.

SECONDARY OUTCOMES:
Comparison with ISHLT classification | 6 months
  • To evaluate the accuracy of INNOGRAFT Heart Suite in discriminating between the classes of rejection according to ISHLT 2004 guidelines using histological study of heart samples from EMB as reference technique
cfDNA modifiers | 6 months
  • To look for potential clinical modifiers of cfDNA levels, as quantitatively determined through INNOGRAFT Heart Suite, for every given rejection class

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Favalli, PhD, Study Director — Myway Gentics Srl
Locations (1):
- IRCCS Fondazione Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Statistical aalysisi will be available at the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR